CLINICAL TRIAL: NCT01479673
Title: Tight Caloric Balance in ICU Patients: a Multicenter, Prospective, Randomized, Controlled Study.
Brief Title: TICACOS International
Acronym: P2 -RMCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Pierre singer, Professor Pierre Singer, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4329
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Mechanical Ventilation Complication
Keywords: Enteral Nutrition; Parenteral Nutrition; Indirect Calorimetry; Intravenous Feeding
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Patients in this group will receive enteral nutrition/parenteral nutrition or combination of enteral and parenteral nutrition according to the "liberal " regimen, i.e. according to local practice.
- Indirect Calorimetry (Experimental): Study group: Indirect Calorimetry (IC) Patients in this group will receive enteral nutrition/parenteral nutrition or combination of enteral and parenteral nutrition according to the individual energy requirements calculated by Indirect Calorimetry measurement of Resting Energy Expenditure (REE).
  Interventions: Dietary Supplement: Indirect Calorimetry measurement of Resting Energy Expenditure .

INTERVENTIONS:
Dietary Supplement: Indirect Calorimetry measurement of Resting Energy Expenditure . — Patients in this group will receive enteral nutrition/parenteral nutrition or combination of enteral and parenteral nutrition according to the individual energy requirements calculated by Indirect Calorimetry.
  Arms: Indirect Calorimetry

SUMMARY:
The aim of this study is to perform a prospective, randomized, controlled blinded study in critically patients to assess the necessity for measuring daily resting energy expenditure as a guide for nutritional support. Our hypothesis is that tight caloric control will reduce the rate of new infections.

Study Design :Multi-center, randomized, single blinded, controlled study. Study Population: newly-admitted, adult mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
Study objectives

To evaluate the effect of tight caloric control in critical patients on:

* The rate of acquired nosocomial infections (Ventilated associated pneumonia, Catheter related infections, Urinary tract infections)
* Mortality rates, length of stay in the ICU and in hospital, length of ventilation and incidence of non-infectious complications.

Primary endpoint:

Rate of nosocomial infections (for definitions see appendage 1) acquired after 48 to 72 hours following admission.

Secondary endpoints

* Metabolic control: glucose concentration, insulin administration, rate of hypoglycemic events.
* Success of tight caloric control: accumulative and maximum negative energy balance.
* Organ function: SOFA score.
* Rate of non-infectious complications: requirement for surgery or occurrence of pressure sores.
* Length of ICU stay and of assisted ventilation (LOS and LOV)
* ICU survival rate.
* Patient status and disposition on day 28 or at hospital discharge.
* 3 & 6 months survival.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically-ventilated adults(Male or Female)admitted to general ICU within the first 48 hours of ICU admission.
2. Age ≥ 18 years;no upper age limit.
3. Expected stay in ICU> 3 days: [SAPS II (18) > ICU median or high-level of nursing care implemented or per clinical impression of attending physician]
4. Medical and abdomino/thoracic surgery patients, as well as multiple trauma patients with Glasgow Coma Score ≥ 10.

Exclusion Criteria:

1. Pregnancy.
2. DNR order.
3. Readmission in the ICU during the same hospitalization/transfer from other ICU.
4. Admission for postoperative monitoring.
5. Respiratory instability: SpO2 <90% or need for ventilator adjustments during the preceding hour or hyperventilation (Respiratory rate > 35/min)
6. Bicarbonate infusion, loss of bicarbonate (diarrhea, ureterosogmoidostomy or use of acetazoloamide, ultrafiltration).
7. Aerosolization with nitric oxide or heliox, tracheal insufflations or visible leaks in chest drainage system.
8. FiO2 80% or patients requiring prone position
9. Chronic/acute liver failure:Child-Pugh class C
10. Brain injury for various reasons with Glasgow Coma Scale below 10.
11. Cardiac surgery patients.
12. Patients in the hospital for more than 7 days.
13. Contra indication to use enteral nutrition.
14. Participation in a clinical study with an investigational drug within one month prior to the start of this clinical trial.
15. Ethical issues that will influence subject eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Rate of nosocomial infections | After 48 to 72 hours /daily assessment: within 28 day
  Rate of nosocomial infections acquired after 48 to 72 hours following admission up to day 28/or discharge will be evaluated

SECONDARY OUTCOMES:
Metabolic control | Day 1 up to day 28/or discharge
  Glucose concentration, insulin administration, rate of hypoglycemic events will be daily assessed
Caloric control | Day 1 up to day 28/or discharge
  Success of tight caloric control:accumulative and maximum negative energy balance

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, MD, Professor, Principal Investigator — RabinMC,Beilinson Hospital; Milana Grinev, RN,Study Coordinator, Study Director — RabinMC, Beilinson Hospital ,Petah- Tikva, Israel
Locations (1):
- Rabin Medical Center, Campus Beilinson, Petah Tikva, Petach Tikva, Israel